CLINICAL TRIAL: NCT03846869
Title: Major Cations Targeted Fluid Therapy In Renal Transplantation.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Marwa Ibrahim Mohamed Abdo,MD, lecturer of anesthesia and surgical intensive care unit principal investigator, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R.19.01.383
Record Dates: First submitted 2019-02-07; First posted 2019-02-20 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Renal Transplant Failure
Keywords: Fluid Therapy; Anesthesia; Renal Transplantation

STUDY DESIGN:
Intervention Model Description: Prospective Cohort Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- major cations (Experimental): bood sample
  Interventions: Diagnostic Test: major cations

INTERVENTIONS:
Diagnostic Test: major cations — blood sample

SUMMARY:
English Summary And Abstract

The overall anesthetic goal for the newly transplanted kidney is to maintain intravascular volume and avoid decreased perfusion by maintaining main arterial blood pressure (MAP). The participants with end-stage renal disease(ESRD) present with electrolyte and metabolic abnormalities such as hyponatremia, hyperchloremia, hyperkalemia, hypocalcemia, hypermagnesemia and metabolic acidosis. With fluid therapy for the participants with (CKD), electrolytes are potentially affected. So there is a progressive metabolic acidosis. The debate about the type of fluid to be used in renal transplant participants is on-going.

Material and methods Place of research is the Department of Anesthesia and Surgical ICU, Urology and Nephrology Center, Faculty of Medicine, Mansoura University, Mansoura, Egypt.Total duration will be assumed to conduct the search over one year. A prospective cohort study and sample size 50 participants aged18 to 40 years. Written informed consent will be obtain from the participants with chronic renal failure scheduled for living-related kidney transplantation surgery .

Basal Serum major cations Na,K,Ca,Mg and Cl, Albumine and after completion of the vascular anastomosis.Fluid therapy volume 40ml/kg From the start of surgery until the renal vessels are unclamped after completion of the vascular anastomosis. and the type of fluid is determined by major cations values. Heart rate ,Systolic, diastolic, mean arterial blood pressure,will be record after induction of anesthesia, every 30 minutes till at the time of renal artery clamping in the donor, at unclamping of the vessels , after completion of the vascular anastomosis and at the end of surgery.the investigator also record renal ischemia time.Time of onset of urine production on unclamping of the renal artery .Total urine output from unclamping of the renal vessels to the end of the surgery.Kidney turgidity will evaluated .

All participants transfer to post-anaesthesia care unit then to ICU .Daily serum creatinine, creatinine clearance, a total urine output and any renal complications will be record for first 5 days postoperatively .

DETAILED DESCRIPTION:
Material and methods Place of research the Department of Anesthesia and Surgical ICU, Urology and Nephrology Center, Faculty of Medicine, Mansoura University, Mansoura, Egypt.

Total duration assumed to conduct the search over one year.

Preoperative management Will be that

* All transplantations in this study will be performed by the same surgical team. All undergo participants preoperative hemodialysis 24 hours before renal transplant surgery.
* Full medical and surgical history will be taken, and
* Routine laboratory investigations (eg. blood Hb, plasma proteins, coagulation studies, serum electrolytes, blood glucose, arterial blood gases, chest radiograph, and echocardiography).
* Basal Serum major cations Na,K,Ca,Mg and Cl, Albumine

Intraoperative management will be

* On the morning of surgery intra muscular injection of Morphine 0.1mg\kg and diclofenac Na 0.6mg/kg. ketamine infusion by rate 0.1 mg /kg/ h
* Monitoring before induction of anesthesia, 5-lead electro cardio gram, pulse oximetry, and noninvasive arterial blood pressure are record. Central venus catheter will be aseptically inserted into the right internal jugular vein ,
* Induction of general anesthesia is with IV midazolam 0.15 mg/kg ,fentanyl 1micogram /kg, and sodium thiopental 5% 5mg/ kg. Endotracheal intubation is facilitated by rocuronium 0.5 mg/kg Anesthesia is maintained by sevoflurane (MAC )minimal alveolar concentration (1%) with 40% O2. Minute volume is adjusted to keep end-tidal CO2approximately 35 mm Hg.
* Fluid therapy volume 40-50 ml/kg From the start of surgery until the renal vessels are unclamped after completion of the vascular anastomosis. and the type of fluid is determined by major cations values.

K > 4.0 ml Eq/dl the investigator use saline 0.9% K<3.5ml Eq/dl us the investigator ringer acetate . k> 5.0ml Eq/dl the investigator use glucose 25% 8gm+ 10 unite insulin in saline 0.9%+salbutamol 200mg.

G Na >140ml Eq/dl the investigator use ringer acetate . Na <135ml Eq/dl the investigator use saline 0.9%. and Na bicarbonate (Na H2CO3) with dose = body weight x base deficit x 0.4 x 1/2

Cl >105 ml Eg/dl the investigator use ringer acetate. Mg<2ml Eq/dl investigator use Mg sulfate 10mg/kg infusion Ca <9ml Eq/dl investigator use Ca gluconate 10% 0.25ml/kg infusion.

* From the start of surgery until the renal vessels are unclamped after completion of the vascular anastomosis. Norepinephrine will infused using infusion pump with started rate 0.01ml/ h and will be adjusted to maintain arterial blood pressure within 25% of the basal value after unclamping at the end of vascular anastomosis or mane arterial blood pressure <60 ml mercury.
* During vascular anastomosis, all recipients will receive 500 mg prednisolone as prepared by the attending nephrologist. After completing the renal vascular anastomosis, furosemide was given in20mg increments to enhance diuresis post vascular anastomosis
* Serum major cations Na,K,Ca,Mg and Cl,Albumine and arterial blood gases will be sampled.
* Heart rate ,Systolic, diastolic, mean arterial blood pressure,will be record after induction of anesthesia, every 30 minutes till at the time of renal artery clamping in the donor(onset of ischemia), at unclamping of the vessels after completion of the vascular anastomosis (end of ischemia),and at the end of surgery.
* The investigator also record renal ischemia time.
* Time of onset of urine production on unclamping of the renal artery in minute.
* Total urine output from unclamping of the renal vessels to the end of the surgery.
* Kidney turgidity will evaluated by the surgical team members, 3-point scale: score I (soft graft), score II (moderate turgid graft), and score III (highly turgid and firm graft).

Post operative management,

* All participants will be assessed for the presence of tissue edema, especially in the conjunctiva, eyelids, face,and upper airway
* All participants had a routine postoperative chest radiograph to look for signs of pulmonary edema and to exclude pneumothorax.
* Daily serum creatinine, creatinine clearance, and total urine output will be record for 5 days postoperatively.
* the investigator also will record any renal complications in the first 5 days (e.g., acute graft rejection, acute tubular necrosis, or need for hemodialysis).

Statistical Analysis

The calculated sample size of the study will be 23 at 5% participants level of significance and 80 % power, using the following formula:

N= (Z1-α/2+Z1-β) ² σ1* σ2 / δ Z1-α/2 = 1.96 Z1-β= 0.842 σ = (Standard deviation δ = Expected difference to be detected between the sample and population α = Level of acceptability of a false positive result (level of significance=0.05) β = Level of acceptability of a false negative result (0.20)

1- β= power (0.80) The sample size will be increased to 50 participants to compensate for drop outs or protocol failures with incomplete data and to increase the study power.

ELIGIBILITY:
Inclusion Criteria:-

- Participants with chronic renal failure scheduled for living-related kidney transplantation surgery

Exclusion Criteria:-

* participants with severe left ventricular dysfunction.
* cardiomyopathy with ejection fraction 50%.
* severe anemia (blood hemoglobin Hb5g\ dL).
* bleeding tendency .
* previously received transplants.
* experienced any surgical complications (e.g., excessive bleeding or resistant graft arterial spasm.
* any surgical difficulty such as the presence of multiple renal vessels.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
normalization acid-base status, intracellular and extracellular water content and plasma electrolyte compositions measured by Serum major cations Na level . | up to 72 weeks
  Serum major cations will be sampled basal and at the time of onset of urine production on unclamping of the renal artery Na ml Eq /dl.
good graft perfusion and early renal function for participants of renal transplantation measured by Total urine output | up to 72 weeks
  Total urine output from de clamping of the renal vessels to the end of the surges in ml
normalization acid-base status, intracellular and extracellular water content and plasma electrolyte compositions measured by Serum major cations K level . | up to 72 weeks
  Serum major cations will be sampled basal and at the time of onset of urine production on unclamping of the renal artery
  ,K ml Eq /dl
normalization acid-base status, intracellular and extracellular water content and plasma electrolyte compositions measured by Serum major cations Ca level. . | up to 72 weeks
  Serum major cations will be sampled basal and at the time of onset of urine production on unclamping of the renal artery
  ,Ca ml Eq /dl
normalization acid-base status, intracellular and extracellular water content and plasma electrolyte compositions measured by Serum major cations Mg levels . | up to 72 weeks
  Serum major cations will be sampled basal and at the time of onset of urine production on unclamping of the renal artery Mg ml Eq /dl.
normalization acid-base status, intracellular and extracellular water content and plasma electrolyte compositions measured by Serum chloride level . | up to 72 weeks
  Serum major cations will be sampled basal and at the time of onset of urine production on unclamping of the renal artery Choride ml Eq /dl
normalization acid-base status, intracellular and extracellular water content and plasma electrolyte compositions measured by Serum albumin level . | up to 72 weeks
  Serum major cations will be sampled basal and at the time of onset of urine production on unclamping of the renal artery Albumin in g
normalization acid-base status, intracellular and extracellular water content and plasma electrolyte compositions measured by arterial blood gases . | up to 72 weeks
  Serum major cations will be sampled basal and at the time of onset of urine production on unclamping of the renal artery arterial blood gases (PH,carbon dioxide partial pressure , bicarbonate ,Base status)
good graft perfusion and early renal function for participants of renal transplantation measured by Total urine output . . | up to 72 weeks
  Total urine output from de clamping of the renal vessels to the end of the surgery in ml
good graft perfusion and early renal function for participants of renal transplantation measured by Kidney turgidity . | up to 72 weeks
  -Kidney turgidity will evaluated by the surgical team members, 3-point scale: score I (soft graft), score II (moderate turgid graft), and score III (highly turgid and firm graft).
good graft perfusion and early renal function for participants of renal transplantation measured by Post operative, Daily serum creatinine, | up to 72 weeks
  -Post operative, Daily serum creatinine,
good graft perfusion and early renal function for participants of renal transplantation measured by Post operative, Daily creatinine clearance . | up to 72 weeks
  Daily creatinine clearance
  .
good graft perfusion and early renal function for participants of renal transplantation measured by total urine output | up to 72 weeks
  total urine output will be recorded for 5 days post operatively in ml

CONTACTS AND LOCATIONS:
Overall Officials: marwa abdo, MD, Principal Investigator — Lecturer of anesthesia and surgical intensive care
Locations (1):
- Marwa Ibrahim Mohamed Abdo, Al Mansurah, Egypt

REFERENCES:
- [Background] Aref A, Zayan T, Sharma A, Halawa A. Utility of central venous pressure measurement in renal transplantation: Is it evidence based? World J Transplant. 2018 Jun 28;8(3):61-67. doi: 10.5500/wjt.v8.i3.61. PMID 29988941
- [Background] Aitken E, Stevenson R, Hanif F, Raj D, Stevenson K, et al. (2016) .Renal Transplantation: An Update for Anaesthetists. Int J Anesthetic Anesthesiol 3:052.
- [Background] Siedlecki A, Irish W, Brennan DC. Delayed graft function in the kidney transplant. Am J Transplant. 2011 Nov;11(11):2279-96. doi: 10.1111/j.1600-6143.2011.03754.x. Epub 2011 Sep 19. PMID 21929642
- [Background] Benjamin S Martinez, Irina Gasanova and Adebola O Adesanya (2013) . Anesthesia for Kidney Transplantation-A ReviewAne. J Anesth Clin Res 4: 2
- [Background] Pfortmueller C, Funk GC, Potura E, Reiterer C, Luf F, Kabon B, Druml W, Fleischmann E, Lindner G. Acetate-buffered crystalloid infusate versus infusion of 0.9% saline and hemodynamic stability in patients undergoing renal transplantation : Prospective, randomized, controlled trial. Wien Klin Wochenschr. 2017 Sep;129(17-18):598-604. doi: 10.1007/s00508-017-1180-4. Epub 2017 Mar 2. PMID 28255797
- [Background] Chaumont M, Racape J, Broeders N, El Mountahi F, Massart A, Baudoux T, Hougardy JM, Mikhalsky D, Hamade A, Le Moine A, Abramowicz D, Vereerstraeten P. Delayed Graft Function in Kidney Transplants: Time Evolution, Role of Acute Rejection, Risk Factors, and Impact on Patient and Graft Outcome. J Transplant. 2015;2015:163757. doi: 10.1155/2015/163757. Epub 2015 Sep 10. PMID 26448870
- [Background] Othman MM, Ismael AZ, Hammouda GE. The impact of timing of maximal crystalloid hydration on early graft function during kidney transplantation. Anesth Analg. 2010 May 1;110(5):1440-6. doi: 10.1213/ANE.0b013e3181d82ca8. PMID 20418304
- [Background] Gezer M, Bulucu F, Ozturk K, Kilic S, Kaldirim U, Eyi YE. Effectiveness of the Stewart Method in the Evaluation of Blood Gas Parameters. Turk J Emerg Med. 2016 Mar 2;15(1):3-7. doi: 10.5505/1304.7361.2014.73604. eCollection 2015 Mar. PMID 27437520
- [Background] Aulakh NK, Garg K, Bose A, Aulakh BS, Chahal HS, Aulakh GS. Influence of hemodynamics and intra-operative hydration on biochemical outcome of renal transplant recipients. J Anaesthesiol Clin Pharmacol. 2015 Apr-Jun;31(2):174-9. doi: 10.4103/0970-9185.155144. PMID 25948896
- [Background] Noritomi DT, Pereira AJ, Bugano DD, Rehder PS, Silva E. Impact of Plasma-Lyte pH 7.4 on acid-base status and hemodynamics in a model of controlled hemorrhagic shock. Clinics (Sao Paulo). 2011;66(11):1969-74. doi: 10.1590/s1807-59322011001100019. PMID 22086530
- [Background] Potura E, Lindner G, Biesenbach P, Funk GC, Reiterer C, Kabon B, Schwarz C, Druml W, Fleischmann E. An acetate-buffered balanced crystalloid versus 0.9% saline in patients with end-stage renal disease undergoing cadaveric renal transplantation: a prospective randomized controlled trial. Anesth Analg. 2015 Jan;120(1):123-129. doi: 10.1213/ANE.0000000000000419. PMID 25185593
- [Background] Schmid S, Jungwirth B. Anaesthesia for renal transplant surgery: an update. Eur J Anaesthesiol. 2012 Dec;29(12):552-8. doi: 10.1097/EJA.0b013e32835925fc. PMID 23010898
- [Background] Yarlagadda SG, Coca SG, Garg AX, Doshi M, Poggio E, Marcus RJ, Parikh CR. Marked variation in the definition and diagnosis of delayed graft function: a systematic review. Nephrol Dial Transplant. 2008 Sep;23(9):2995-3003. doi: 10.1093/ndt/gfn158. Epub 2008 Apr 11. PMID 18408075
- [Background] Toth M, Reti V, Gondos T. Effect of recipients' peri-operative parameters on the outcome of kidney transplantation. Clin Transplant. 1998 Dec;12(6):511-7. PMID 9850443
- [Background] Baxi V, Jain A, Dasgupta D. Anaesthesia for renal transplantation: an update. Indian J Anaesth. 2009 Apr;53(2):139-47. PMID 20640114
- [Background] Yee J, Parasuraman R, Narins RG. Selective review of key perioperative renal-electrolyte disturbances in chronic renal failure patients. Chest. 1999 May;115(5 Suppl):149S-157S. doi: 10.1378/chest.115.suppl_2.149s. PMID 10331349